CLINICAL TRIAL: NCT05924659
Title: Evaluation of Neurofeedback Training's Efficiency for the Optimization of Attentionnal Performances
Brief Title: Neurofeedback Training's Efficiency for Attentionnal Performances
Acronym: ENOCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Collaborators: Hotel Dieu de France Hospital (Other); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023_ENOCA; 2022-A02306-37 (Other: IDRCB)
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Attention-deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized assigment, neurofeedback training versus control
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double bling computizded neurofeed back training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback Training (Experimental): 1 week of cerebral training with a neurofeedback strategy based on increased alpha EEG activity
  Interventions: Other: Cerabral training
- Control (Sham Comparator): 1 week of cerebral training with a strategy based on time on task increase of performance, without neurofeedback
  Interventions: Other: Cerabral training

INTERVENTIONS:
Other: Cerabral training — 1 week of cerebral training (neurofeedback or sham)

SUMMARY:
This randomised, double bling and controled study aim to evaluate the performance of a neurofeedback training on attentional capabilities, in comparison to placebo. We hypothesize 1) that an electroencephalographic (EEG) based neurofeedback training may improve attentional performances of healthy subjects, and 2) inter-individual variability might be explained by factors such as body awarness, sleep parameters and genetics of individuals.

DETAILED DESCRIPTION:
Many jobs require high attentional performances that are maintained over time, which imply safety issues. Just like physicial performances of top athletes, it is possible to use a set of innovative methods and technologies to improve cognitive performances (attention, working memory, decision making… ), in particular with the help of brain training programs such as neurofeedback protocoles. Although neurofeedback training efficiency has been evaluated in many context (either with patients or healthy subjects), it is still a subject of debate. More specifically, inter-individual variability is far from beeing understood. We hypothesize 1) that an electroencephalographic (EEG) based neurofeedback training may improve attentional performances of healthy subjects, and 2) inter-individual variability might be explained by factors such as body awarness, sleep parameters and genetics of individuals.

1. To demonstrate the efficiency of EEG neurofeedback (EEG-NFB) trainings versus a control group, we will compare the conflict monitoring score obtained with the Attentional Network Task (Reaction Times (RT) in ms of Incongruent trials minus Reaction Times of Congruent trials : RTincongruent - Rtcongruent). Our hypothesis is a reduction of the conflict monitoring scores after the EEG-NFB compared to baseline (before EEG-NFB), and a lower score for the EEG-NFB group compared to the control group.
2. To describe the different factors influencing EEG-NFB training efficacy, we will explore the inter-individual variability by assessing the body awarness (especially cardiac interoceptive accuracy with a counting task), sleep parameters (hypnogram, sleep power spectral activities) and genetic polymorphisms (DRD2, COMT, DAT1, PER3, ADA, ADORA2A, TNF-α).

The study design will be a controlled interventional protocol, double-blinded with parralel-arms (EEG-NFB vs Control) in healthy volunteers.

* Prior informations will be given to individuals expressing an interest in this study.
* During the inclusion, an investigator or a member of the research team will verbally reiterate the informations and answer any additional questions. The volunteer will be reminded of his/her rights in the contexte of research involving the human person.
* After verifying volunteer's eligibility criteria, he/she will be asked to sign the consent form.
* Volunteers will have to fill out a sleep questionnaire.Sleep/wake cycles will be home monitored with a wearable headset during 14 days : 7 days before the start of EEG-NFB training, and 7 during the EEG-NFB training.
* Cognitive tests will be done each day of EEG-NFB training (or control) : Psychomotor Vigilance Task, Attentional Network Test, AX-Continuous Performance Test and a Heartbit Counting task. The cognitive test period will last 30 minutes.
* EEG-NFB training (or control) will be done for 5 consecutive days, each session lasts 35 min (10 blocs of 3 min, and short breaks of 30 s). Each session will be precedeed and followed by a resting-state recording. The control group will perform a SHAM EEG-NFB.
* Before the first session and after the last (5th) session, cortisol and α-amylase concentrations will be evaluated by saliva tests.
* Before the session and after the last session, questionnaires evaluating body awarness will be filled out by volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female volunteers
* aged between 18 yo and 50 yo.

Exclusion Criteria:

* any pathological issues,
* previous traumatic brain and/or auditive injuries,
* volunteers having already experienced NFB trainings,
* high tobacco consumers,
* volunteers refusing genotyping.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Attentional performance | One week
  the Attentional Network Task (Reaction Times (RT) in ms of Incongruent trials minus Reaction Times of Congruent trials : RTincongruent - Rtcongruent).

SECONDARY OUTCOMES:
Sleep parameters | One week
  Total sleep duration in minutes

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut de recherche biomédicale des armées, Brétigny-sur-Orge
  - Hotel Dieu, Paris

IPD SHARING:
Plan to Share IPD: No